CLINICAL TRIAL: NCT05804721
Title: Comparative Randomized, Single Dose, Two-way Crossover Bioequivalence Study to Determine the Bioequivalence Aripiprazole From Apipe 10 mg Orally Disintegrating Tablets (Man. by: P&C Labs (Pellets & CR Products), Egypt) Versus Abilify 10 mg Orodispersible Tablets (Otsuka Pharmaceutical Netherlands B.V., Netherlands)
Brief Title: Bioequivalence Study of Aripiprazole From Apipe 10 mg Orally Disintegrating Tablets (Man. by: P&C Labs (Pellets & CR Products), Egypt) Versus Abilify 10 mg Orodispersible Tablets (Otsuka Pharmaceutical Netherlands B.V., Netherlands)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: P&C Labs, Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/22/1016
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T test (Experimental): 1 orally disintegrating tablet contains 10 mg Aripiprazole administrated according to a randomization scheme with 240 ml of water
  Interventions: Drug: Apipe (Aripiprazole10 mg)
- R Reference (Active Comparator): 1 orodispersible tablet contains 10 mg Aripiprazole administrated according to a randomization scheme with 240 ml of water
  Interventions: Drug: Abilify (Aripiprazole10 mg)

INTERVENTIONS:
Drug: Apipe (Aripiprazole10 mg) — Test drug
  Other Names: Abilify
  Arms: T test
Drug: Abilify (Aripiprazole10 mg) — Reference drug
  Other Names: Abilify
  Arms: R Reference

SUMMARY:
Comparative randomized, single dose, two-way crossover bioequivalence study to determine the bioequivalence of Aripiprazole from Apipe 10 mg orally disintegrating tablets (Man. by: P&C Labs (Pellets&CR Products), Egypt) versus Abilify 10 mg orodispersible tablets (Otsuka Pharmaceutical Netherlands B.V., Netherlands ) in Healthy Human Volunteers Under Fasting Condition

DETAILED DESCRIPTION:
Healthy male volunteers, 45-55 years of age, selected from the Egyptian population fulfilling the selection criteria. 24 subjects will participate in the study. All dosed subject samples will be analyzed and their data will be included in the final study report 18 blood samples will be drawn in each period. The total volume of blood will not exceed 200 ml throughout the whole study. 0.00, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00 hours.

Primary Pharmacokinetic Parameters: Cmax, Truncated AUC0→72 Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax and Truncated AUC0→72 for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios for Truncated AUC0→72 and Cmax to be within 80.00-125.00%.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, age 45 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Fully informed subjects that consented to participate in the study.
6. Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

1. Females
2. Subjects with a prior personal or family history of dystonic reactions to medications.
3. Subjects with known allergy or any contraindications to the products tested.
4. Heavy smokers (more than 10 cigarettes per day).
5. Subjects that do not agree not to consume alcohol-containing beverages and foods for 48 hours before dosing and throughout the period of sample collection
6. Subjects whose values of BMI were outside the accepted normal ranges.
7. Medical demographics with evidence of clinically significant deviation from normal medical condition.
8. Results of laboratory tests which are clinically significant.
9. Acute infection within one week preceding first study drug administration.
10. History of drug or alcohol abuse.
11. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
12. Subject is on a special diet (for example subject is vegetarian).
13. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
14. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
15. Subject has a history of severe diseases which have direct impact on the study.
16. Participation in a bioequivalence study or in a clinical study within the last 8 weeks before first study drug administration.
17. Subject intends to be hospitalized within 3 months after first study drug administration.
18. Subjects who have blood donated or lost more than 500 mL blood within 3 months prior to the study.

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 72 hours post dose in each treatment period
  to measure the maximal measured plasma concentration

SECONDARY OUTCOMES:
Tmax | Up to 72 hours post dose in each treatment period
  time of the maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861